CLINICAL TRIAL: NCT02093715
Title: FeNO and Cytokines in RSV and Non RSV Bronchiolitis in Relation to Future Asthma
Brief Title: FeNO and Cytokines in Respiratory Syncytial Virus (RSV) and Non RSV Bronchiolitis in Relation to Future Asthma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-13-YS-07-075-CTIL
Record Dates: First submitted 2014-03-19; First posted 2014-03-21 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-06

CONDITIONS: Acute Bronchiolitis
Keywords: Bronchiolitis; FeNO; Asthma; wheezing, RSV
MeSH Terms: conditions — Bronchiolitis; Asthma; Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Biospecimen Retention: Samples Without DNA — blood

GROUPS / COHORTS (5):
- RSV: Infant with acute bronchiolitis due to RSV
- Co- Infection: Infant with acute bronchiolitis due to RSV and other respiratory virus
- Other: Infant with acute bronchiolitis due to non-RSV respiratory virus
- Unknown: Infant with acute bronchiolitis with negative PCR results for respiratory viruses
- Control: Healthy infants

SUMMARY:
The purpose of this study is to determine Fractional exhaled Nitric-Oxide (FeNO)levels and blood cytokines during acute bronchiolitis, and to seek for correlation between these markers and future development of asthma.

ELIGIBILITY:
Inclusion Criteria:

* First episode of shortness of breath
* Children in ages 2 weeks to 2 years

Exclusion Criteria:

* Any chronic disease
* Congenital anomalies

Ages: 2 Weeks to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children ages 2 weeks to 2 years who will arrive to Dana Children's hospital, Tel-Aviv Medical Center due to first episode of shortness of breath and working diagnosis of bronchiolitis.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2007-07; Primary Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Physician diagnosed asthma | At the age of 4 years
  Modification of The International Study of Asthma and Allergies in Childhood (ISAAC) questionnaires

SECONDARY OUTCOMES:
Fractional exhaled Nitric Oxide (FENO) level | During acute bronchiolitis, after 2 and 6 months
  FeNO level measured by a rapid-response chemiluminescence analyzer (Eco Physics CLD88 NO analyzer, EcoMedics AG,Switzerland).

OTHER OUTCOMES:
Wheezing episode | From recruitment time till the age 4.
PCR for respiratory viruses | At recruitment
  Polymerase chain reaction (PCR) analysis of nasal secretion for: RSV, Influenza A, Influenza B, Pandemic H1N1, Adenovirus, human metapneumovirus (hMPV), Parainfluenza 1-3, Enterovirus, Bocavirus, Rhinovirus, Corona virus-229E, Corona-OC43, Corona-HKU1 and Corona-NL63.

CONTACTS AND LOCATIONS:
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel